CLINICAL TRIAL: NCT06425562
Title: The Potential Added Value of Impulse Oscillometry in Asthma Monitoring
Acronym: AM-IOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24151_AM-IOS
Record Dates: First submitted 2024-04-30; First posted 2024-05-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: impulse oscillometry; asthma monitoring
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult asthma patients (Experimental): Lung function tests (full lung function, multiple breath nitrogen washout, impulse oscillometry) and questionaires (asthma control test, asthma control questionnaire, asthma quality of life questionnaire) will be conducted, once at baseline and once 3 - 6 months later during follow-up.
  Interventions: Other: Full lung function; Other: Multiple breath nitrogen washout; Other: Impulse oscillometry

INTERVENTIONS:
Other: Full lung function — This includes spirometry, body plethysmography and single breath gas transfer test. These are all non-invasive physiological measurements / lung function tests. Measures flow volumes, lung volumes and gas transfer respectively.
Other: Multiple breath nitrogen washout — Non-invasive physiological measurement / lung function test. 100% oxygen is inhaled and the nitrogen concentration in the lungs is measured. This test gives information on the ventilation distribution in the lungs.
Other: Impulse oscillometry — Non-invasive physiological measurement / lung function test. This technique superimposes sound waves on tidal breathing. The patient can breathe normally trough the device, no forced respiratory maneuvers are required. It gives information on the reactance and resistance of the lung.

SUMMARY:
The goal of this longitudinal observational study is to learn if impulse oscillometry (IOS) has an added value in asthma monitoring in adult asthma patients who are prescribed a change in asthma maintenance therapy. The main questions it aims to answer are:

* Is there a difference in the change in IOS parameters and FEV1 respectively, stratified according to change in asthma control test?
* Is there a difference in the change in IOS parameters and FEV1 respectively, stratified according to change in other questionnaire such as the asthma control questionnaire and the asthma quality of life questionnaire.
* Are the proposed minimal clinically important differences (MCIDs) valid for short follow-up periods (3 - 6 months)?

Participants will undergo lung function testing (full lung function, multiple breath nitrogen washout, impulse oscillometry) and questionnaires (asthma control test, asthma control questionnaire, asthma quality of life questionnaire), once during the baseline visit and once during the follow-up visit three to six months later.

ELIGIBILITY:
Inclusion Criteria:

* Adult asthma patients with a scheduled consultation at the outpatient hospital to whom a step-up or step-down of their pharmacological asthma treatment is prescribed

Exclusion Criteria:

* Unstable asthma (defined as need for oral corticosteroids or (respiratory) antibiotic course in the 4 weeks before inclusion or any major medical issue in the 4 weeks before inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in frequency dependance of resistance (FDR) stratified according to change in asthma control test (ACT) | Once at baseline and 3 - 6 months later during follow-up
  Frequency dependance of resistance (FDR) is an impulse oscillometry parameter. FDR is expressed in kPa/(L.s). A lower FDR indicates a clinically better outcome. The ACT is a questionnaire which consists of 5 questions, each evaluated on a 5-point Likert-Scale. Total score ranges between 5 and 25, where a lower score is clinically worse than a higher score.
Change in area of reactance (AX) stratified according to change in asthma control test (ACT) | Once at baseline and 3 - 6 months later during follow-up
  Area of reactance (AX) is an impulse oscillometry parameter. AX is expressed in kPa/L. A lower AX indicates a clinically better outcome. The ACT is a questionnaire which consists of 5 questions, each evaluated on a 5-point Likert-Scale. Total score ranges between 5 and 25, where a lower score is clinically worse than a higher score.
Change in forced expiratory volume in 1 second (FEV1) stratified according to change in asthma control test (ACT) | Once at baseline and 3 - 6 months later during follow-up
  Spirometry parameter: forced expiratory volume in 1 second (FEV1). FEV1 is expressed in L. A higher FEV1 indicates a clinically better outcome. The ACT is a questionnaire which consists of 5 questions, each evaluated on a 5-point Likert-Scale. Total score ranges between 5 and 25, where a lower score is clinically worse than a higher score.

SECONDARY OUTCOMES:
Change in frequency dependence of resistance (FDR) stratified according to change in asthma control questionnaire (ACQ-6) | Once at baseline and 3 - 6 months later during follow-up
  Frequency dependance of resistance (FDR) is an impulse oscillometry parameter. FDR is expressed in kPa/(L.s). A lower FDR indicates a clinically better outcome. The ACQ-6 is a questionnaire which consists of 6 questions, each evaluated on a 7-point Likert-Scale. The total score score is divided by 6 yielding a mean score ranging from 0.0 to 6.0, where a lower score is clinically better than a higher score.
Change in area of reactance (AX) stratified according to change in asthma control questionnaire (ACQ-6) | Once at baseline and 3 - 6 months later during follow-up
  Area of reactance (AX) is an impulse oscillometry parameter. AX is expressed in kPa/L. A lower AX indicates a clinically better outcome. The ACQ-6 is a questionnaire which consists of 6 questions, each evaluated on a 7-point Likert-Scale. The total score score is divided by 6 yielding a mean score ranging from 0.0 to 6.0, where a lower score is clinically better than a higher score.
Change in forced expiratory volume in 1 second (FEV1) stratified according to change in asthma control questionnaire (ACQ-6) | Once at baseline and 3 - 6 months later during follow-up
  Spirometry parameter: forced expiratory volume in 1 second (FEV1). FEV1 is expressed in L. A higher FEV1 indicates a clinically better outcome. The ACQ-6 is a questionnaire which consists of 6 questions, each evaluated on a 7-point Likert-Scale. The total score score is divided by 6 yielding a mean score ranging from 0.0 to 6.0, where a lower score is clinically better than a higher score.
Change in frequency dependence of resistance (FDR) stratified according to change in asthma quality of life questionnaire (AQLQ) | Once at baseline and 3 - 6 months later during follow-up
  Frequency dependance of resistance (FDR) is an impulse oscillometry parameter. FDR is expressed in kPa/(L.s). A lower FDR indicates a clinically better outcome. The AQLQ is a questionnaire which consists of 32 questions, each evaluated on a 7-point Likert-Scale. The total score is divided by 32 yielding a mean score ranging from 1.0 to 7.0, where a lower score is clinically worse than a higher score.
Change in area of reactance (AX) stratified according to change in asthma quality of life questionnaire (AQLQ) | Once at baseline and 3 - 6 months later during follow-up
  Area of reactance (AX) is an impulse oscillometry parameter. AX is expressed in kPa/L. A lower AX indicates a clinically better outcome.The AQLQ is a questionnaire which consists of 32 questions, each evaluated on a 7-point Likert-Scale. The total score is divided by 32 yielding a mean score ranging from 1.0 to 7.0, where a lower score is clinically worse than a higher score.
Change in forced expiratory volume in 1 second (FEV1) stratified according to change in asthma quality of life questionnaire (AQLQ) | Once at baseline and 3 - 6 months later during follow-up
  Spirometry parameter: forced expiratory volume in 1 second (FEV1). FEV1 is expressed in L. A higher FEV1 indicates a clinically better outcome.The AQLQ is a questionnaire which consists of 32 questions, each evaluated on a 7-point Likert-Scale. The total score is divided by 32 yielding a mean score ranging from 1.0 to 7.0, where a lower score is clinically worse than a higher score.
Change in frequency dependence of resistance (FDR) over the 3-6 months observation period compared to proposed minimal clinically important differences (MCIDs) (calculated for a one year interval) for FDR. | Once at baseline and 3 - 6 months later during follow-up
  MCIDs over 1 year have been published for IOS parameters. For frequency dependence of resistance (FDR) the MCID is defined as a decline of FDR greater or equal to 0.06 kPa/(L.s). Change of FDR ≥ 0.06 kPa/(L.s) or not
Change in area of reactance (AX) over the 3-6 months observation period compared to proposed minimal clinically important differences (MCIDs) (calculated for a one year interval) for AX. | Once at baseline and 3 - 6 months later during follow-up
  MCIDs over 1 year have been published for IOS parameters. For area of reactance (AX) the MCID is defined as a decline of AX greater or equal to 0.65 kPa/L. Change of AX ≥ 0.65 kPa/L or not

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No